CLINICAL TRIAL: NCT06823999
Title: Effect of Vitamin C in the Prevention and Treatment for Bruises in Patients with Ischemic Stroke: a Double-blind Randomized Control Trial
Brief Title: Prevention and Treatment for Bruises in Patients with Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2024099
Record Dates: First submitted 2025-01-20; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Bruises; Skin Lesions
Keywords: stroke; bruises; skin lesions; vitamin C; bleeding
MeSH Terms: conditions — Stroke; Contusions; Hemorrhage | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stroke (Experimental)
  Interventions: Drug: Ascorbic acid (Vitamin C)
- Control (Placebo Comparator): Participants receiving normal saline 20 ml infusion perday for 4 days
  Interventions: Other: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Ascorbic acid (Vitamin C) — In the study, acute ischemic stroke patients will receiving vitamin C 4 gram perday for 4 days.
  Arms: stroke
Other: Normal Saline (Placebo) — Particiapnts receiving normal saline 20 ml perday for 4 days
  Arms: Control

SUMMARY:
Background Over the past few decades, significant advances have been made in the diagnosis and treatment of strokes. Most studies focus on functional recovery in stroke patients. In addition to motor function, there are many symptoms may affect function and quality of life in stroke patients. Bruises are caused by damage to the skin that causes blood to drain out of the capillaries and accumulate in the connective tissue of the skin or subcutaneous tissue. The study on non-motor syndrome in ischemic stroke patients found that 25.8% of ischemic stroke patients had bruises and 17.7% of bruises were unexplained bruises. In addition to the physiological and emotional effects on stroke patients, bruises may increase infection risk and affect stroke patient outcomes. Vitamin C is a natural antioxidant discovered in 1747 to treat and prevent scurvy. Vitamin C can reduce gum bleeding and prevent colon bleeding after a polypectomy. Vitamin C has been reported to reduce brain edema around brain injury and decrease mortality in patients with traumatic brain injury. Dehydroascorbic acid decreases infarct volume in mice with middle cerebral artery occlusion. Investigators hypothesized that administration of vitamin C to patients with acute ischemic stroke patients would decrease the risk of bleeding and enhance its resolution. Investigators also hypothesized that vitamin C injection could minimize infarct volume and improve outcomes in ischemic stroke patients. The aims of the study include: 1. To investigate whether vitamin C injections can reduce bruising risk and enhance bruising resolution. 2. To explore whether vitamin C injections in the acute phase of stroke can improve the prognosis of ischemic stroke patients.

Methods This is a prospective, double-blind, randomized controlled study. All patients admitted to the hospital under the diagnosis of ischemic stroke and stroke was confirmed by Magnetic Resonance imaging (MRI) or brain computed imaging (CT) and aged between 20 and 85 years were invited to participate in the study. Investigators excluded patients who had these diseases: cancer receiving chemotherapy, end stage renal disease receiving dialysis, autoimmune disease, hematological disease, Glucose-6-phosphatase disease, gouty arthritis, and a lack of informed consent.

During the study period, all patients who met the inclusion and exclusion criteria were invited to participate in the study. After informed consent, participants were randomly assigned to the experimental group or the control group. All participants underwent NIHSS evaluation and a detailed dermatological examination on the day of hospitalization. After enrollment, the experimental group received 4 mg Vitamin C injection per day for 4 days, while the control group received the same volume of normal saline injection per day for 4 days. Researchers evaluate participant skin condition (including bruises number and size, color) every day during hospitalization, and up to 1 month after stroke. Investigators evaluate NIHSS at discharge and follow-up functional outcome (mRS) up to 3 months after stroke onset.

Analysis Rate shows bruise percentage. Chi square or Fisher exact test was applied to compare the difference in bruises between two groups. Logistic regression was used to compare bruise risk between groups. Wilcoxon rank sign test was used to analyze stroke severity and outcome between two groups.

DETAILED DESCRIPTION:
Introduction

Background Stroke is one of the most severe diseases that causes mortality and morbidity. With the latest advances in stroke prevention and treatment, stroke incidence and mortality have significantly reduced. Advances in imaging technology have improved ischemic stroke diagnosis. The establishment of a stroke center and the improvement of procedures will allow stroke patients to be treated faster. Advances in medical technology include advances in imaging technology, endovascular thrombectomy(1, 2), and advances in pharmaceuticals include tissue plasminogen activator(3), anticoagulant(4), and antiplatelet drugs(5) lead to better outcomes for stroke patients. Current research on stroke focuses on motor function treatment. However, besides reduced limb strength, stroke patients still have many symptoms that deserve attention. Although these diseases do not directly affect motor function, they will cause physical and psychological obstacles and affect stroke patients' quality of life. For example, depression, post-stroke pain, sleep disorders, bedsores, bruises, and infection, are all common problems after a stroke and deserve attention. In addition to limb weakness in stroke patients, the occurrence of the above-mentioned conditions will prolong hospitalization time, increase hospitalization expenses, and affect treatment results. The more common problems are post-infarction bleeding, infection, and stroke. Stroke patients also often suffer from non-neurological complications, which affect patient treatment outcomes and neurological recovery (6). Common complications include cardiovascular diseases, pulmonary embolism, sleep disorders, pain, falls, venous thrombosis, infections, and bleeding. Bruising is an often- clinical issue caused by blood leaking from blood vessels and accumulating in the tissue beneath the skin. The most common cause of bruising is blunt force trauma, which leads to subcutaneous vascular rupture and blood leakage. Other common causes include drug injections, the underlying disease, or treatment for the disease. Age is also a factor influencing bruising. In elderly individuals, skin degeneration results in a thinner epidermis, fragile blood vessels, and reduced subcutaneous tissue, making them more prone to bruising (7).

Elderly patients often have more medical conditions, increasing bruising. Medications such as antithrombotic and anticoagulant drugs also heighten bruising risk. Bruising can also result from vitamin deficiencies (8). Although most bruises fade over time, with color changing during the process, the timing of the bruise cannot be accurately determined by color changes, as the rate of resolution varies among individuals (9). However, bruises may sometimes indicate more severe underlying conditions (10).

For instance, abdominal bruising found might be a sign of internal bleeding. Bruising around the mastoid region or behind the ear may indicate skull fractures. Bruising in the scrotum, perineum, or anterior abdomen wall may suggest abdominal aortic rupture (11). In addition to being associated with severe diseases, bruising also increases infection risk and affects patient recovery (12).

If bruising is observed in children, especially in those who are not capable of moving on their own, abuse should be considered. Research indicates that bruising in infants is a potential marker of abuse and warrants attention. While the causes of bruises in older adults differ from those in children, unexplained bruising in the elderly also requires investigation, as elder abuse remains a concern. Bruising in older individuals may also be the result of abuse (13).

The hospital's research team found that 25.8% of stroke patients exhibit bruising. This is with 55.4% of cases occurring before hospitalization and 44.6% during hospitalization. Of these, 17.7% of bruises are unknown. These unexplained bruises could be due to minor injuries that patients are unaware of, concealment, abuse, other underlying diseases, or medication-related causes, all of which merit further investigation.

However, beyond investigating bruising causes, the most crucial steps are to treat existing bruises and prevent further occurrences. Previous research on bruising focuses on its prevention and treatment after surgery. To date, there is still no simple and effective method to prevent bruising (14).

Vitamin C is a natural vitamin. As early as 1747, the connection between scurvy and vitamin C was suspected and the first use of a randomized controlled trial was conducted to study this relationship. In the experiment, 12 scurvy patients were divided into two groups: six in the experimental group consumed foods high in vitamin C, while the control group did not. The results showed that scurvy patients who consumed vitamin C-rich foods recovered quickly, while those who did not showed no improvement.

Vitamin C is an essential cofactor for enzymes and a powerful antioxidant. It plays a critical role in synthesizing neurotransmitters, collagen, and maintaining endothelial cell function (15). An adult non-smoker typically has about 1.5 grams of vitamin C in their body, consuming about 60 milligrams daily. Smokers consume more vitamin C, approximately 140 milligrams per day. In cases of illness, such as surgery, trauma, infection, or shock, blood levels of vitamin C drop rapidly, requiring supplementation through injection (16).

Stroke patients have lower vitamin C blood concentrations than healthy individuals. Vitamin C protects neurons and reduces ischemic damage.

Vitamin C protects blood vessels. Research indicates that in patients undergoing colorectal polyp removal, administering 500 mg of vitamin C two hours before the procedure significantly reduces the post-polypectomy bleeding rate (17).

A comprehensive study found that supplementing vitamin C in individuals with low blood levels reduces the incidence of gum bleeding and retinal hemorrhages (18). Previous research showed that administering high doses of vitamin C to patients with severe brain injuries decreases the extent of brain edema around the injury site and lowers mortality rates (19).

Previous studies demonstrated that high-dose vitamin C enhances critically ill patients' response to vasopressors, preserves endothelial barrier function, prevents cell apoptosis, and increases recovery rates after cardiopulmonary resuscitation in critically ill patients (20). However, other studies have shown that while high-dose vitamin C in sepsis patients reduces vasopressor use and the rate of acute organ failure, it does not lower mortality rates (21).

A study found that patients with atrophic gastritis who took high doses of vitamin C (500 mg daily) over an extended period, compared to those taking 50 mg daily, had significantly reduced levels of reactive oxygen species (ROS), which are aging and cancer-inducing factors, in their blood (22). Long-term use of vitamin C reduces oxidative stress, decreases protein aggregation in the brain, and may help mitigate neurodegenerative diseases.

Vitamin C is a safe and inexpensive medication, and it is safe beyond doubt. In an animal study by Judy et al., it was found that in rats experiencing middle cerebral artery occlusion followed by reperfusion, administering oxidized vitamin C reduced the infarct size by 53% to 59% (23). In an animal experiment, rats were subjected to middle cerebral artery occlusion for 60 minutes, followed by reperfusion for 30 or 60 minutes. Rats injected with vitamin C had higher blood levels of Ten eleven translocase and 5-hydroxymethylcytosine than those not injected with vitamin C, and the infarct size was smaller (24). Stroke patients aged 65 and older with higher blood concentrations of vitamin C had a 50% reduced mortality rate than those with low concentrations (25). In comparison to healthy adults, stroke patients had lower blood concentrations of vitamin C, and increased levels of inflammatory markers (CRP, ICAM-1, MCP-1), and increased oxidative stress (8-epiPGF2), indicating an inflammatory response in stroke patients (26). A meta-analysis found that individuals who consumed more vitamin C and had higher blood concentrations of vitamin C had a lower risk of stroke (27).

Based on previous research showing that high-dose vitamin C injections can decrease bleeding rates during colorectal polyp removal (17) and decrease the incidence of gum and retinal bleeding (18), the first hypothesis of this study is that vitamin C has a protective effect on blood vessels. It may aid in vascular repair, reduce bruising, and accelerate bruise recovery. Since high-dose vitamin C has been shown to reduce brain ischemia (15, 28), the second hypothesis is that acute stroke patients have low blood vitamin C levels. Vitamin C injections can improve micro-vascular blood flow in the brain, aiding stroke patients' recovery (29).

Beyond its visual impact, bruising can also affect psychologically (30), increase the risk of infection, influence patient outcomes (12, 31), and impact physicians' medication choices. Currently, there is limited research on bruising in stroke patients, and few studies explore the relationship between vitamin C and ischemic stroke. This study aims to enhance understanding of the impact of bruising in stroke patients, its prevention and treatment, and the effects of vitamin C on stroke outcomes.

Methods This study was approved by the Institutional Review Board (IRB) of Chia Yi Christian Hospital (Approval Number: IRB2024099). The research subjects were ischemic stroke patients at Chia Yi Christian Hospital.

A. Study Design: This study adopted a parallel design, enrolling hospitalized ischemic stroke patients confirmed by computed tomography (CT) or magnetic resonance imaging (MRI). Patients meeting any exclusion criteria for the study were not included. During the study, participants could withdraw at any time upon request. If adverse drug reactions occurred during the study, the principal investigator could terminate the patient's participation.

To investigate the incidence, causes, and impact of hematoma on stroke patients' treatment outcomes, this study observed and recorded the timing, quantity, resolution time, and resolution rate of hematoma. In addition, it recorded its causes. To explore whether hematoma occurrence could be reduced and recovery accelerated, and to improve stroke patients' treatment outcomes, a double-blind, randomized study design was used. This study focuses on bleeding issues related to stroke patients. It explores the causes and impacts of bruising on treatment outcomes and stroke recurrence, and examines methods of bruising prevention and treatment.

B. Randomized Assignment Randomization was conducted using the National Cancer Institute Clinical Trial Tool (NIH > National Cancer Institute Clinical Trial Tool). Participants were randomly assigned to either the experimental or the control group. The experimental group received daily injections of 4 grams of vitamin C, while the control group received injections of an equivalent volume of normal saline.

C. Participants:

1. Number of Participants (Sample Size):

   The sample size was estimated using G-power. With an alpha error of 0.05, a power of 0.95, and an effect size of 0.2, at least 314 participants were required. This study plans to recruit 400 participants, with 200 in the experimental group and 200 in the control group.

   The evaluation metric is the occurrence of newly formed hematomas during hospitalization.
2. Recruitment of Potential Participants (Target Population, Methods, Locations, etc.):

The recruitment target comprises patients with acute ischemic stroke. Physicians and research assistants from the research team will explain the study's purpose and methods to patients on the stroke ward. Upon consent, the study will proceed.

E. Implementation Methods:

1. The execution process:

   After confirmation of ischemic stroke via computed tomography (CT) or magnetic resonance imaging (MRI), patients meeting the inclusion criteria and willing to participate will be included in the study.

   Participant assessment
   1. Initial Evaluation: Each participant will undergo an assessment of stroke severity (NIHSS) during hospitalization. The NIHSS score is defined as the sum of 15 individually evaluated elements. The NIHSS ranges from 0 to 42. Stroke severity was categorized as follows: 0, no stroke symptoms; 1-4, minor stroke; 5-15, moderate stroke; 16-20, moderate to severe stroke; and 21-42, severe stroke.

      Participants will also undergo a detailed skin evaluation.
   2. Treatment: All participants will receive standard stroke treatment. The experimental group will receive intravenous injections of 4 grams of vitamin C daily for 4 days.

   The control group will receive equivalent volumes of normal saline. Nursing staff will administer injections. The saline solution will be packaged and prepared to match the vitamin C injections in appearance and volume. Dispensing will be done by the clinical trial pharmacy.
2. Follow-Up and Necessary Care Plan for Participants:

   Researchers will assess participants' bruise development and recovery progress during hospitalization and after discharge until three weeks after stroke onset. Researchers will assess participants' functional abilities for up to 3 months.

   For unexplained hematomas, necessary diagnostic tests will be performed to investigate potential underlying diseases.
3. Primary and Secondary Outcomes:

O Primary Outcomes:

1. The rate of hematoma occurrence (in any location) up to 2 weeks post-stroke. 2. Comparison of hematoma resolution rates up to 3 weeks post-stroke, using a benchmark of a reduction in hematoma area greater than 30%. This applies to both pre-existing and newly developed hematomas.

O Secondary Outcomes:

1. Changes in stroke severity, comparing NIHSS scores at admission and discharge. This will evaluate whether vitamin C injections reduce post-stroke neurological deterioration. A NIHSS increase of more than 3 is considered neurological deterioration.
2. Functional outcomes at three months post-stroke, measured using the Modified Rankin Scale (mRS). A mRS do not exceeding 2 is considered a good outcome, and a mRS exceeding 2 is considered a poor outcome.
3. Investigation of hematoma causes, including exploration of whether hematomas indicate other underlying conditions.

O Safety Outcomes:

1. Evaluation of vitamin C injection safety, including adverse reaction monitoring.
2. In cases of adverse drug reactions, the principal investigator will assess whether to terminate the patient's participation in the study.

3 Random Allocation Table. After the patient signs the consent form, participants will be grouped according to the severity of the stroke.

The groups are divided into two based on stroke severity: one group includes 200 participants with mild strokes (NIHSS 0-4) and one group includes participants with NIHSS 5-20.

Participants in treatment

1. Preparation of medication:

   Research Assistant (A) prepares the list of medications needed for the day and organizes the required injections.

   Based on the patient's group assignment, the medication is provided to the attending nurse, who administers the injection.
2. Skin and Hematoma Assessment:

Research Assistant (B) collaborates with the nurse to assess the patient's skin condition, recording and photographing any hematomas present.

The skin and hematoma condition will be monitored and tracked for one month post-discharge.

Statistical analysis

1. Descriptive Statistics: Percentages will be used to describe bruising occurrence rates and the causes of different types of bruising.

   Bruising will be calculated in terms of days before and after hospitalization. An analysis of the bruises will be presented as counts and percentages. Broken rates in different age groups will be shown as percentages. Bruising resolution rates will be presented in days. The bleeding area will be estimated using square centimeters, and changes will be compared. A reduction of 30% in the bruising area after 4 days of treatment will be considered a response.

   This method will be used for presenting the main outcomes. Differences between the two groups will be compared using the Chi-square test.
2. Inferential Statistics: For normally distributed continuous data, the mean ± standard deviation (mean ± SD) will be applied; for non-normally distributed data, the median will be applied. Normally distributed data will be compared using a T-test (e.g., age, PT, PTT, INR). Non-normally distributed data (e.g., NIHSS, mRS) will be compared using the Mann-Whitney U test.

For categorical variables, differences will be assessed using the Chi-square or Fisher exact test (e.g., diabetes, hypertension, hyperlipidemia, and other stroke risk factors).

Logistic regression will be used for multivariable analysis. (3) Period Analysis: A mid-term analysis will be conducted at the end of the first year.

Expected tasks to be completed

1. Understand the prevalence of bruising in stroke patients and its impact on them.
2. Clearly identify the causes of bruising and explore the proportion associated with medications or medical interventions.
3. Understand the psychological and physiological effects of bruising on stroke patients.
4. Determine if high-dose vitamin C injections can reduce bruising in stroke patients and promote early resolution.
5. Clearly assess the impact of high-dose vitamin C injections on ischemic stroke treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke patients.
* Aged 20 to 85 years.

Exclusion Criteria:

* o Cancer patients undergoing chemotherapy.

  * End-stage renal disease patients receiving hemodialysis.
  * Patients undergoing immunosuppressive therapy.
  * Patients with coagulation disorders.
  * Patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency (favism).
  * Patients with thalassemia.
  * Patients who did not sign the consent form.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — No special selection.
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
1. The rate of hematoma occurrence (in any location). 2. Comparison of hematoma resolution rates, using a benchmark of a reduction in hematoma area greater than 30%. This applies to both pre-existing and newly developed hematomas. | The study will begin at Auguest 1, 2025, we evaluate patients skin condition everyday and analysis the results at August 2027.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarraj A, Hassan AE, Abraham MG, Ortega-Gutierrez S, Kasner SE, Hussain MS, Chen M, Blackburn S, Sitton CW, Churilov L, Sundararajan S, Hu YC, Herial NA, Jabbour P, Gibson D, Wallace AN, Arenillas JF, Tsai JP, Budzik RF, Hicks WJ, Kozak O, Yan B, Cordato DJ, Manning NW, Parsons MW, Hanel RA, Aghaebrahim AN, Wu TY, Cardona-Portela P, Perez de la Ossa N, Schaafsma JD, Blasco J, Sangha N, Warach S, Gandhi CD, Kleinig TJ, Sahlein D, Elijovich L, Tekle W, Samaniego EA, Maali L, Abdulrazzak MA, Psychogios MN, Shuaib A, Pujara DK, Shaker F, Johns H, Sharma G, Yogendrakumar V, Ng FC, Rahbar MH, Cai C, Lavori P, Hamilton S, Nguyen T, Fifi JT, Davis S, Wechsler L, Pereira VM, Lansberg MG, Hill MD, Grotta JC, Ribo M, Campbell BC, Albers GW; SELECT2 Investigators. Trial of Endovascular Thrombectomy for Large Ischemic Strokes. N Engl J Med. 2023 Apr 6;388(14):1259-1271. doi: 10.1056/NEJMoa2214403. Epub 2023 Feb 10. PMID 36762865
- [Background] Veunac L, Saliou G, Knebel JF, Bartolini B, Puccinelli F, Michel P, Hajdu SD. Revascularization of carotid artery occlusion using stenting versus non stenting in endovascular management of tandem occlusion stroke. J Clin Neurosci. 2022 Apr;98:15-20. doi: 10.1016/j.jocn.2022.01.036. Epub 2022 Feb 4. PMID 35131720
- [Background] Hacke W, Kaste M, Fieschi C, von Kummer R, Davalos A, Meier D, Larrue V, Bluhmki E, Davis S, Donnan G, Schneider D, Diez-Tejedor E, Trouillas P. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Second European-Australasian Acute Stroke Study Investigators. Lancet. 1998 Oct 17;352(9136):1245-51. doi: 10.1016/s0140-6736(98)08020-9. PMID 9788453
- [Background] Essebag V, Healey JS, Joza J, Nery PB, Kalfon E, Leiria TLL, Verma A, Ayala-Paredes F, Coutu B, Sumner GL, Becker G, Philippon F, Eikelboom J, Sandhu RK, Sapp J, Leather R, Yung D, Thibault B, Simpson CS, Ahmad K, Toal S, Sturmer M, Kavanagh K, Crystal E, Wells GA, Krahn AD, Birnie DH. Effect of Direct Oral Anticoagulants, Warfarin, and Antiplatelet Agents on Risk of Device Pocket Hematoma: Combined Analysis of BRUISE CONTROL 1 and 2. Circ Arrhythm Electrophysiol. 2019 Oct;12(10):e007545. doi: 10.1161/CIRCEP.119.007545. Epub 2019 Oct 15. PMID 31610718
- [Background] Johnston SC, Easton JD, Farrant M, Barsan W, Conwit RA, Elm JJ, Kim AS, Lindblad AS, Palesch YY; Clinical Research Collaboration, Neurological Emergencies Treatment Trials Network, and the POINT Investigators. Clopidogrel and Aspirin in Acute Ischemic Stroke and High-Risk TIA. N Engl J Med. 2018 Jul 19;379(3):215-225. doi: 10.1056/NEJMoa1800410. Epub 2018 May 16. PMID 29766750
- [Background] Kumar S, Selim MH, Caplan LR. Medical complications after stroke. Lancet Neurol. 2010 Jan;9(1):105-18. doi: 10.1016/S1474-4422(09)70266-2. PMID 20083041
- [Background] Sinikumpu SP, Jokelainen J, Haarala AK, Keranen MH, Keinanen-Kiukaanniemi S, Huilaja L. The High Prevalence of Skin Diseases in Adults Aged 70 and Older. J Am Geriatr Soc. 2020 Nov;68(11):2565-2571. doi: 10.1111/jgs.16706. Epub 2020 Aug 4. PMID 32754902
- [Background] Pahadiya HR, Lakhotia M, Choudhary S, Prajapati GR, Pradhan S. Reversible ecchymosis and hyperpigmented lesions: A rare presentation of dietary Vitamin B12 deficiency. J Family Med Prim Care. 2016 Apr-Jun;5(2):485-487. doi: 10.4103/2249-4863.192343. PMID 27843871
- [Background] Mosqueda L, Burnight K, Liao S. The life cycle of bruises in older adults. J Am Geriatr Soc. 2005 Aug;53(8):1339-43. doi: 10.1111/j.1532-5415.2005.53406.x. PMID 16078959
- [Background] Csizmar CM, Abraham HM, Thompson CA. 84-Year-Old Female With Easy Bruising. Mayo Clin Proc. 2023 Jul;98(7):1079-1084. doi: 10.1016/j.mayocp.2022.12.022. Epub 2023 Jun 7. No abstract available. PMID 37278679
- [Background] Epperla N, Mazza JJ, Yale SH. A Review of Clinical Signs Related to Ecchymosis. WMJ. 2015 Apr;114(2):61-5. PMID 26756058
- [Background] Gleva MJ, Poole JE. BRUISE CONTROL INFECTION Study: Blood and Bugs. J Am Coll Cardiol. 2016 Mar 22;67(11):1309-11. doi: 10.1016/j.jacc.2016.01.033. No abstract available. PMID 26988952
- [Background] Wiglesworth A, Austin R, Corona M, Schneider D, Liao S, Gibbs L, Mosqueda L. Bruising as a marker of physical elder abuse. J Am Geriatr Soc. 2009 Jul;57(7):1191-6. doi: 10.1111/j.1532-5415.2009.02330.x. Epub 2009 Jun 3. PMID 19558476
- [Background] Chan DS, Roskies M, Jooya AA, Samaha M. Postoperative Ecchymosis and Edema After Creation of Subperiosteal Tunnels in Rhinoplasty: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2019 Mar 1;21(2):133-136. doi: 10.1001/jamafacial.2018.1716. PMID 30589927
- [Background] Dresen E, Lee ZY, Hill A, Notz Q, Patel JJ, Stoppe C. History of scurvy and use of vitamin C in critical illness: A narrative review. Nutr Clin Pract. 2023 Feb;38(1):46-54. doi: 10.1002/ncp.10914. Epub 2022 Sep 25. PMID 36156315
- [Background] Berger MM. Vitamin C requirements in parenteral nutrition. Gastroenterology. 2009 Nov;137(5 Suppl):S70-8. doi: 10.1053/j.gastro.2009.08.012. PMID 19874953
- [Background] Vahdat Shariatpanahi Z, Shahbazi S, Shahbazi E. Ascorbic Acid to Prevent Postpolypectomy Bleeding in the Colon: A Randomized Controlled Trial. Asian J Endosc Surg. 2022 Jan;15(1):103-109. doi: 10.1111/ases.12977. Epub 2021 Aug 27. PMID 34448547
- [Background] Hujoel PP, Kato T, Hujoel IA, Hujoel MLA. Bleeding tendency and ascorbic acid requirements: systematic review and meta-analysis of clinical trials. Nutr Rev. 2021 Aug 9;79(9):964-975. doi: 10.1093/nutrit/nuaa115. PMID 33517432
- [Background] Razmkon A, Sadidi A, Sherafat-Kazemzadeh E, Mehrafshan A, Jamali M, Malekpour B, Saghafinia M. Administration of vitamin C and vitamin E in severe head injury: a randomized double-blind controlled trial. Clin Neurosurg. 2011;58:133-7. doi: 10.1227/neu.0b013e3182279a8f. No abstract available. PMID 21916138
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Sato R, Hasegawa D, Prasitlumkum N, Ueoka M, Nishida K, Takahashi K, Nasu M, Dugar S. Effect of IV High-Dose Vitamin C on Mortality in Patients With Sepsis: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Crit Care Med. 2021 Dec 1;49(12):2121-2130. doi: 10.1097/CCM.0000000000005263. PMID 34495877
- [Background] Sasazuki S, Hayashi T, Nakachi K, Sasaki S, Tsubono Y, Okubo S, Hayashi M, Tsugane S. Protective effect of vitamin C on oxidative stress: a randomized controlled trial. Int J Vitam Nutr Res. 2008 May;78(3):121-8. doi: 10.1024/0300-9831.78.3.121. PMID 19003734
- [Background] Huang J, Agus DB, Winfree CJ, Kiss S, Mack WJ, McTaggart RA, Choudhri TF, Kim LJ, Mocco J, Pinsky DJ, Fox WD, Israel RJ, Boyd TA, Golde DW, Connolly ES Jr. Dehydroascorbic acid, a blood-brain barrier transportable form of vitamin C, mediates potent cerebroprotection in experimental stroke. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11720-4. doi: 10.1073/pnas.171325998. PMID 11573006
- [Background] Moskowitz A, Huang DT, Hou PC, Gong J, Doshi PB, Grossestreuer AV, Andersen LW, Ngo L, Sherwin RL, Berg KM, Chase M, Cocchi MN, McCannon JB, Hershey M, Hilewitz A, Korotun M, Becker LB, Otero RM, Uduman J, Sen A, Donnino MW; ACTS Clinical Trial Investigators. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Organ Injury in Septic Shock: The ACTS Randomized Clinical Trial. JAMA. 2020 Aug 18;324(7):642-650. doi: 10.1001/jama.2020.11946. PMID 32809003
- [Background] Gale CR, Martyn CN, Winter PD, Cooper C. Vitamin C and risk of death from stroke and coronary heart disease in cohort of elderly people. BMJ. 1995 Jun 17;310(6994):1563-6. doi: 10.1136/bmj.310.6994.1563. PMID 7787644
- [Background] Sanchez-Moreno C, Dashe JF, Scott T, Thaler D, Folstein MF, Martin A. Decreased levels of plasma vitamin C and increased concentrations of inflammatory and oxidative stress markers after stroke. Stroke. 2004 Jan;35(1):163-8. doi: 10.1161/01.STR.0000105391.62306.2E. Epub 2003 Dec 11. PMID 14671251
- [Background] Chen GC, Lu DB, Pang Z, Liu QF. Vitamin C intake, circulating vitamin C and risk of stroke: a meta-analysis of prospective studies. J Am Heart Assoc. 2013 Nov 27;2(6):e000329. doi: 10.1161/JAHA.113.000329. PMID 24284213
- [Background] Morris-Blanco KC, Chokkalla AK, Kim T, Bhatula S, Bertogliat MJ, Gaillard AB, Vemuganti R. High-Dose Vitamin C Prevents Secondary Brain Damage After Stroke via Epigenetic Reprogramming of Neuroprotective Genes. Transl Stroke Res. 2022 Dec;13(6):1017-1036. doi: 10.1007/s12975-022-01007-6. Epub 2022 Mar 20. PMID 35306630
- [Background] Barak OF, Caljkusic K, Hoiland RL, Ainslie PN, Thom SR, Yang M, Jovanov P, Dujic Z. Differential influence of vitamin C on the peripheral and cerebral circulation after diving and exposure to hyperoxia. Am J Physiol Regul Integr Comp Physiol. 2018 Oct 1;315(4):R759-R767. doi: 10.1152/ajpregu.00412.2017. Epub 2018 Jul 11. PMID 29995458
- [Background] Gisondi P, Puig L, Richard MA, Paul C, Nijsten T, Taieb C, Stratigos A, Trakatelli M, Salavastru C; EADV Burden of Skin Diseases Project Team. Quality of life and stigmatization in people with skin diseases in Europe: A large survey from the 'burden of skin diseases' EADV project. J Eur Acad Dermatol Venereol. 2023 Oct;37 Suppl 7:6-14. doi: 10.1111/jdv.18917. PMID 37806002
- [Background] Feldman KW, Tayama TM, Strickler LE, Johnson LA, Kolhatkar G, DeRidder CA, Matthews DC, Sidbury R, Taylor JA. A Prospective Study of the Causes of Bruises in Premobile Infants. Pediatr Emerg Care. 2020 Feb;36(2):e43-e49. doi: 10.1097/PEC.0000000000001311. PMID 29040244